CLINICAL TRIAL: NCT07171801
Title: 3D vs. 2D Unilateral Biportal Endoscopic Spine Surgery: A Randomized Blinded Crossover Pilot Simulation Study
Brief Title: Comparing 3D and 2D Views in Biportal Spine Surgery: A Pilot Simulation Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Felix Corr (Other)
Responsible Party: Sponsor-Investigator, Felix Corr, Stefan Motov, Cantonal Hospital of St. Gallen
Organization: Cantonal Hospital of St. Gallen (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Device Feasibility
Other Study IDs: V1
Record Dates: First submitted 2025-09-06; First posted 2025-09-15 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Spinal Diseases; Endoscopy Simulation; Lumbar Vertebrae; Randomized Controlled Trial; Three-Dimensional; Simulation Training
MeSH Terms: conditions — Spinal Diseases

STUDY DESIGN:
Intervention Model Description: This study employs a randomized, single-center, blinded, crossover design in a high-fidelity simulated surgical environment. Each participant performs standardized unilateral biportal endoscopic spine surgery tasks using both 2D and 3D visualization systems in a randomized sequence. A washout period is incorporated between conditions to minimize carryover effects. This within-subjects crossover model allows each participant to serve as their own control, increasing statistical power and reducing inter-individual variability. Blinding is maintained for performance assessors, and objective motion tracking metrics are used to evaluate technical performance under each visualization condition.
Who Masked: Outcomes Assessor
Masking Description: In this single-center crossover simulation study, outcomes assessors responsible for performance evaluation and motion data analysis are blinded to the visualization modality used during each session (3D or 2D). Participants are not blinded due to the inherent perceptual differences between the two visualization systems. Investigators supervising the simulation are aware of the intervention assignments for operational purposes but are not involved in outcome assessment. All video and motion tracking data are anonymized and coded prior to analysis to maintain assessor blinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Three-Dimensional Endoscopy First, Then Two-Dimensional (Other): Participants first perform standardized spinal endoscopic simulation tasks using a stereoscopic three-dimensional (3D) endoscopic system providing binocular depth perception via dual optical channels and polarized glasses. After completing all tasks under 3D visualization, the same participants subsequently repeat the identical tasks using conventional two-dimensional (2D) visualization on the same high-definition endoscopic platform
  Interventions: Device: Three-Dimensional Endoscopic Visualization; Device: Two-Dimensional Endoscopic Visualization
- Two-Dimensional Endoscopy First, Then Three-Dimensional (Other): Participants first perform standardized spinal endoscopic simulation tasks using conventional two-dimensional (2D) visualization, with stereoscopic capability deactivated, displaying a monoscopic high-definition image. After completing all tasks under 2D visualization, the same participants subsequently repeat the identical tasks using stereoscopic three-dimensional (3D) visualization on the same endoscopic platform, viewed with polarized glasses.
  Interventions: Device: Three-Dimensional Endoscopic Visualization; Device: Two-Dimensional Endoscopic Visualization

INTERVENTIONS:
Device: Three-Dimensional Endoscopic Visualization — Use of a stereoscopic 3D high-definition endoscopic system with dual optical channels, projecting to a stereoscopic monitor viewed with polarized glasses, to perform standardized spinal simulation tasks.
Device: Two-Dimensional Endoscopic Visualization — Use of the same high-definition endoscopic system with stereoscopic function deactivated, providing conventional monoscopic two-dimensional visualization, to perform standardized spinal simulation tasks.

SUMMARY:
This study aims to compare three-dimensional (3D) and two-dimensional (2D) visualization in biportal endoscopic spine surgery using a simulated environment. Surgeons will perform standardized tasks on a spine model while using either 3D or 2D endoscopic systems. The goal is to determine whether 3D technology can improve precision, efficiency, and movement control during surgery. The study uses a randomized, blinded, crossover design to ensure objective results and may help guide future training and technology use in spinal endoscopy.

DETAILED DESCRIPTION:
Spinal endoscopy, particularly the unilateral biportal endoscopic (UBE) technique, is an increasingly adopted minimally invasive approach for treating lumbar spine pathologies. While it offers clinical advantages over traditional open surgery-including less tissue disruption, reduced blood loss, and faster recovery-its uptake has been limited, in part due to the technical challenges associated with two-dimensional (2D) endoscopic visualization. The lack of depth perception inherent to 2D imaging can impair spatial orientation, hand-eye coordination, and surgical precision, especially in anatomically complex regions such as the lumbar spine.

Three-dimensional (3D) endoscopic systems are designed to address this limitation by restoring binocular depth cues and providing stereoscopic visualization. Preliminary evidence from other surgical fields-such as laparoscopy and cranial neurosurgery-suggests that 3D visualization improves operative performance, task efficiency, and user confidence. However, the benefits of 3D visualization in spinal endoscopy remain poorly understood, with no rigorous controlled studies to date assessing its impact on performance metrics under standardized conditions.

This randomized, blinded, crossover pilot study is designed to objectively evaluate the effect of 3D versus 2D endoscopic visualization on technical performance during simulated UBE procedures. Participants-including surgeons at various experience levels-will complete standardized surgical tasks on high-fidelity lumbar spine models using both 2D and 3D endoscopic systems. Motion tracking technology will be employed to quantitatively analyze instrument movement, capturing key metrics such as path length, velocity, motion economy, and high-velocity excursions.

The crossover design ensures that each participant serves as their own control, and blinding minimizes observational bias during performance assessment. The simulation setting allows for reproducible conditions free from patient-related variability, ensuring that observed differences can be attributed to visualization modality rather than anatomical or clinical complexity.

Findings from this study will provide foundational data on the potential utility of 3D visualization in spinal endoscopy, with implications for surgical training, operative safety, and the future integration of stereoscopic technologies in spine surgery.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in the neurosurgical residency or fellowship program at the Department of Neurosurgery, Cantonal Hospital of St. Gallen, Switzerland
* Completion of basic neurosurgical training modules, including introductory endoscopic handling
* Age ≥ 18 years
* Willingness and ability to provide informed consent

Exclusion Criteria:

* Prior substantial experience with three-dimensional (3D) endoscopy (defined as > 5 independent procedures performed with 3D visualization systems)
* Ocular or neurological conditions impairing stereopsis, fine motor control, or safe endoscope handling
* Inability or unwillingness to complete the simulation protocol
* Declined participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Difference in Task Completion Time (seconds) and Error Rate During Spinal Endoscopic Simulation, Assessed Immediately Post-Task | Immediately during each simulation session (within minutes of task performance).
  Task performance was assessed during standardized spinal endoscopic simulation tasks under both three-dimensional (3D) and two-dimensional (2D) visualization. Task completion time was measured in seconds with a digital stopwatch from the start to the successful completion of each task. Task accuracy was assessed as the number of predefined errors, including deviations from the optimal trajectory or inadvertent contact with marked "no-go" zones on the simulation model. Both measures were collected immediately during each simulation session. Lower times and fewer errors indicate better performance.
Difference in Task Completion Time (seconds) and Error Rate During Spinal Endoscopic Simulation, Assessed Immediately Post-Task | Immediately during each simulation session (within minutes of task performance).
  Task performance was assessed during standardized spinal endoscopic simulation tasks under both three-dimensional (3D) and two-dimensional (2D) visualization. Task completion time was measured in seconds with a digital stopwatch from the start to the successful completion of each task. Task accuracy was assessed as the number of predefined errors, including deviations from the optimal trajectory or inadvertent contact with marked "no-go" zones on the simulation model. Both measures were collected immediately during each simulation session. Lower times and fewer errors indicate better performanc

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Motov, MD, Principal Investigator — Kantonsspital St. Gallen, Health Ostschweiz

IPD SHARING:
Plan to Share IPD: No
The study generated only simulation performance and questionnaire data from healthy volunteer trainees. No clinical or patient-level data were collected. Individual-level data will not be shared, but summary results are available in the publication.

REFERENCES:
- [Background] Ban Y, Mcneely B, Chadha NK, Felton M. Safety and efficacy of three-dimensional versus two-dimensional endoscopy in otolaryngology surgery and training: A systematic review. Clin Otolaryngol. 2024 Sep;49(5):538-551. doi: 10.1111/coa.14171. Epub 2024 May 12. PMID 38735751
- [Background] Heo DH, Kim JY, Park JY, Kim JS, Kim HS, Roh J, Park CK, Chung H. Clinical Experiences of 3-Dimensional Biportal Endoscopic Spine Surgery for Lumbar Degenerative Disease. Oper Neurosurg. 2022 Apr 1;22(4):231-238. doi: 10.1227/ONS.0000000000000090. PMID 35147593
- [Background] Ma A, Xie N, Reidy J, Mobbs RJ. Three-dimensional endoscopy in lumbar spine surgery as a novel approach for degenerative pathologies: a case report. J Surg Case Rep. 2024 Aug 28;2024(8):rjae540. doi: 10.1093/jscr/rjae540. eCollection 2024 Aug. PMID 39211372